CLINICAL TRIAL: NCT02208063
Title: A Phase 3 Multicenter, Randomized, Open-label, Clinical Trial of Telavancin Versus Standard Intravenous Therapy in the Treatment of Subjects With Staphylococcus Aureus Bacteremia Including Infective Endocarditis
Brief Title: A Phase 3 Telavancin Staphylococcus Aureus (S. Aureus) Bacteremia Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Halted due to lack of statistical power. No safety concerns identified.
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0112
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Bacteremia
Keywords: Bacteremia; Staphylococcus aureus
MeSH Terms: conditions — Bacteremia; Staphylococcal Infections | interventions — telavancin; Vancomycin; Daptomycin; Nafcillin; Oxacillin; Cloxacillin; Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telavancin (Experimental): 7.5 mg/kg administered intravenously once every 24 hours daily over 60 minutes
  Interventions: Drug: Telavancin
- Standard of care (Active Comparator): Vancomycin, Daptomycin, synthetic penicillin or Cefazolin
  Interventions: Drug: Vancomycin; Drug: Daptomycin; Drug: Synthetic penicillin; Drug: Cefazolin

INTERVENTIONS:
Drug: Telavancin
  Arms: Telavancin
Drug: Vancomycin
  Arms: Standard of care
Drug: Daptomycin
  Other Names: Cubicin
  Arms: Standard of care
Drug: Synthetic penicillin
  Other Names: Nafcillin; Oxacillin; Cloxacillin
  Arms: Standard of care
Drug: Cefazolin
  Arms: Standard of care

SUMMARY:
This is a multicenter, randomized, open-label, noninferiority trial of telavancin versus standard IV therapy control (e.g., vancomycin, daptomycin, anti-staphylococcal penicillin (PCN), or cefazolin) in the treatment of subjects with complicated Staphylococcus aureus (S. aureus) bacteremia and SA right-sided infective endocarditis (SA-RIE).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with at least one blood culture positive for S. aureus within 48 hours before randomization
* At least one of the following signs or symptoms of bacteremia:

  * Temperature ≥ 38.0°C
  * White blood cell (WBC) count > 10,000 or < 4,000 cells/µL or > 10% immature neutrophils (bands)
  * Tachycardia (heart rate > 90 bpm)
  * Tachypnea (respiratory rate > 20 breaths/min)
  * Hypotension (systolic blood pressure < 90 mmHg)
  * Signs or symptoms of localized catheter-related infection
* At enrollment, subjects must have either 1) known right-sided infective endocarditis by Modified Duke's criteria 2) known complicated bacteremia, demonstrated as signs or symptoms of metastatic foci of S. aureus infection or 3) at least one risk factor for complicated bacteremia.

Exclusion Criteria:

* Treatment with any potentially effective (anti-staphylococcal) systemic antibiotic for more than 60 hours within 7 days before randomization. EXCEPTION: Documented resistance to the prior systemic antibacterial therapy
* Presence of an infection source that will not be managed or controlled within the first 3 days of study drug treatment
* Presence of prosthetic cardiac valve or cardiac device (eg, implantable cardioverter defibrillator [ICD]), permanent pacemaker, or cardiac valve support ring)
* Known or suspected left-sided infective endocarditis (LIE), by Modified Duke Criteria. NOTE: Right-sided infective endocarditis (RIE) is permitted
* Known or suspected osteomyelitis or meningitis. NOTE: Evidence of metastatic complications related to the primary infection such as right-sided endocarditis, septic arthritis, septic pulmonary emboli are permitted. S. aureus pneumonia is permitted
* Confirmed evidence (identification or gram stain) of a mixed polymicrobial infection with a Gram-negative pathogen that requires non-study antibiotic treatment with agent(s) that have activity against Gram-negative pathogens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (1):
- Remington-Davis Clinical Research, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Telavancin: 7.5 mg/kg administered intravenously once every 24 hours daily over 60 minutes
  Telavancin
- Standard of Care: Vancomycin, Daptomycin, synthetic penicillin or Cefazolin
  Vancomycin
  Daptomycin
  Synthetic penicillin
  Cefazolin
Period: Overall Study
Arm/Group | Telavancin | Standard of Care
Started (All Randomized) | 60 | 61
Randomized and Treated | 58 | 60
Microbiological All Treated (Includes all subjects in the AT population who had a mono-microbial QBC positive for S. aureus.) | 47 | 52
Completed | 48 | 50
Not Completed | 12 | 11
Not completed — Death | 3 | 5
Not completed — Not Specified in report | 3 | 4
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic (All-Treated Population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Telavancin | Standard of Care | Total
Number analyzed (Participants) | 57 | 60 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (16.41) | 56.5 (16.33) | 54.5 (16.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 39 | 43 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 19 | 39
  Not Hispanic or Latino | 37 | 41 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Black or African American | 8 | 5 | 13
  White | 44 | 48 | 92
  Other | 2 | 2 | 4
  Missing | 0 | 1 | 1
  Multiple | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinical Outcome of Cure at Test of Cure (TOC)
Description: The efficacy endpoint of clinical outcome of cure at the test of cure (TOC) was determined by subjects who meet all of the following criteria, as determined by the investigator and adjudicated by the blinded independent efficacy adjudication committee (IEAC).
  1. Alive at TOC
  2. Resolution of all clinical signed and symptoms of the Staphylococcus aureus (S. aureus) infection at TOC
  3. No evidence of microbiological persistence of relapse
  4. No new foci of metastatic S. aureus infection after Day 8
Time Frame: Up to 8 weeks
Population: One subject enrolled was excluded from all summaries and analyses because the subject was randomized to a higher dose of telavancin (10mg/kg) that the remainder of the subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Telavancin | Standard of Care
Number analyzed (Participants) | 47 | 52
Participants
  Cure | 22 | 27
  Failure | 19 | 21
  Indeterminate | 6 | 4

2. Secondary Outcome: Number of Participants With an Investigator Clinical Outcome of Cure at TOC in the Microbiological All-treated (mAT) Population
Description: The efficacy endpoint of Investigator clinical outcome of cure at the test of cure (TOC) was determined by the following criteria:
  1. Subject alive at TOC
  2. Resolution of all clinical signs and symptoms of the S. aureus infection at TOC (unless explained by a more likely alternative diagnosis)
  3. No evidence of microbiological persistence or relapse
  4. No new foci of metastatic S. aureus infection after Day 8
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Telavancin | Standard of Care
Number analyzed (Participants) | 47 | 52
Participants
  Cure | 26 | 31
  Failure | 15 | 19
  Indeterminate | 3 | 0
  Missing | 3 | 2

3. Secondary Outcome: Investigator Clinical Response (Success or Failure) at EOT in the Microbiological All-treated (mAT) Population
Description: This efficacy endpoint was determined to be a clinical failure if the subject switched study antibiotic due to lack of clinical response
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Telavancin | Standard of Care
Number analyzed (Participants) | 47 | 52
Participants
  Success | 28 | 36
  Failure | 13 | 15
  Indeterminate | 5 | 0
  Missing | 1 | 1

4. Secondary Outcome: Number of Participants With the Development of a New Metastatic Foci of S. Aureus Infection at Test of Cure (TOC) in the Microbiological All-treated (mAT) Populations
Description: After Day 8, any sign or symptom leading to a subsequent confirmed diagnosis of a new metastatic foci of S. aureus infection
Time Frame: Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Telavancin | Standard of Care
Number analyzed (Participants) | 47 | 52
Participants
  Yes | 6 | 3
  No | 32 | 41
  Indeterminate | 9 | 8

ADVERSE EVENTS:
Time Frame: 38 months
Arm/Group | Telavancin | Standard of Care
All-Cause Mortality (participants affected / at risk) | 3/58 | 5/60
Serious Adverse Events (participants affected / at risk) | 16/58 | 13/60
Other Adverse Events (participants affected / at risk) | 29/58 | 25/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telavancin (N=58) | Standard of Care (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Unintentional medical device removal (General disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Serratia infection (Infections and infestations) | 1 (1) | 0 (0)
Spinal empyema (Infections and infestations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telavancin (N=58) | Standard of Care (N=60)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 7 (7)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Constipation (Gastrointestinal disorders) | 3 (3) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (10) | 8 (8)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 8 (8)

LIMITATIONS AND CAVEATS:
At the interim analysis, study was deemed to be inadequately powered & terminated prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT02208063/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT02208063/SAP_001.pdf